CLINICAL TRIAL: NCT03886298
Title: For Patients With Pancreatic Cancer Pain, Does Radiofrequency Splanchnic Denervation Isprovide a Similar Analgesia as Neurolytic Celiac Block
Brief Title: Radiofrequency Splanchnic Denervation Versus Retrocrural Neurolytic Celiac Block for Pancreatic Cancer Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Diab Fuad Hetta, Principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SECI-IRB-IORG0009563-725
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radiofrequency splanchnic denervation (Experimental)
  Interventions: Procedure: radiofrequency splanchnic denervation
- retrocrural celiac denervation (Active Comparator)
  Interventions: Procedure: retrocrural celiac denervation

INTERVENTIONS:
Procedure: radiofrequency splanchnic denervation — the authors will denervate the splanchnic nerves via radiofrequency
  Arms: radiofrequency splanchnic denervation
Procedure: retrocrural celiac denervation — the authors will denervate the splanchnic nerves in the retrocrural space via injection of alcohol
  Arms: retrocrural celiac denervation

SUMMARY:
The investigators will evaluate the analgesic efficacy of radiofrequency splanchnic nerve denervation versus neurolytic retrocrural celiac denervation for patients with abdominal pain due to cancer pancreas

ELIGIBILITY:
Inclusion Criteria:

* patients with abdominal pain due to cancer pancreas

Exclusion Criteria:

* coagulopathy
* infection at site of the procedure

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-04-10 (Estimated); Study Completion 2020-06-10 (Estimated)

PRIMARY OUTCOMES:
the percentage of patients that gain more than 50% reduction of their pain on VAS pain score | 6 months postoperatively
  VAS pain scale is a tool for measurement of pain intensity scored from 0 to 10 in which 0 + no pain and 10 + the worst pain immaginable

CONTACTS AND LOCATIONS:
Locations (1):
- Diab, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided